CLINICAL TRIAL: NCT04044365
Title: Development and Psychometric Testing of a Pediatric Chronic Graft- Versus-Host Disease (GVHD) Symptom Scale (PCSS)
Brief Title: Pediatric cGVHD Symptom Scale
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190131; 19-C-0131
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12-09

CONDITIONS: Graft vs Host Disease
Keywords: Hematopoietic Stem Cell Transplantation (HSCT); Allogeneic Stem Cell Transplant; Phototherapies; Graft Vs Host Disease; Natural History
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 1/Project 1 Child/caregiver-proxy: Children age 5-7 with cGVHD and their caregiver, n=20 child/parent dyads
- 2/Project 1 Child/caregiver-proxy: Children age 8-12 with cGVHD and their caregiver, n=35 child/parent pairs
- 3/Project 1 Child/caregiver-proxy: Children age 13-17 with cGVHD and their caregiver, n=35 child/parent pairs
- 4/Project 2 Child/caregiver-proxy: Children age 5-7 with cGVHD and their caregiver, n=40 child/parent pairs
- 5/Project 2 Child/caregiver-proxy: Children age 8-12 with cGVHD and their caregiver, n=40 child/parent pairs
- 6/Project 2 Child/caregiver-proxy: Children age 13-17 with cGVHD and their caregiver, n=40 child/parent pairs

SUMMARY:
Background:

Some children/adolescents who have had a stem cell transplant live with chronic graft-versus-host-disease (cGVHD). cGVHD is a side effect of the transplant that can cause multiple bothersome symptoms and negatively affect a child/adolescent squality of daily life. The questionnaires that measure thesymptoms caused by cGVHD are designed for adults. Children/adolescents may not describe their symptoms in the same way. The goal of this research is to improve the way we measure how bothersome these symptoms are for children/adolescents living with cGVHD.

Objective:

To develop a questionnaire (The Pediatric cGHVD Symptom Scale) for children/adolescents living with cGVHD to identify the symptoms they are experiencing and describe how bothersome those symptoms are to them. An additional goal is to design a parent/guardian companion questionnaire that can be used to capture the symptom experiences of very young children who may not be able to complete a questionnaire.

Eligibility:

Children/adolescents ages 5-17 who are receiving treatment for cGVHD after a stem cell transplant, and their parent/guardian..

Design:

This study consists of 2 projects.

Children/adolescents with cGVHD and their parent/guardianparticipants will be grouped by the child/adolescent s age: 5-7, 8-12, and 13-17.

In project 1, participants will complete an age-appropriate questionnaire about cGVHD symptoms. The questionnaire will ask about the child/adolescent s physical functioning and emotional well-being. The parent/guardian will out fill out a companion questionnaire online. The child/adolescent will then review their completed questionnaire during an interview with a researcher and will be asked whether the questions about their symptoms were difficult to understand. The parent/guardian and child/adolescent will then be interviewed together to further explore their responses to the questionnaires. Interviews will be done in person, by phone, and online. . Based on what is learned through these interviews, the wording of the questionnaire will be improved for better comprehension and ease of response.

In project 2, participants will complete this revised questionnairefor their age group along with some other questionnaires that ask about quality of life. Both the child/adolescent and parent/guardian will fill out the questionnaires online at three separate time points.

In both projects, children/adolescents with cGVHD and their parent/guardian participants will be grouped by the child/adolescent s age: 5-7, 8-12, and 13-17.

...

DETAILED DESCRIPTION:
Background:

* Hematopoietic stem cell transplantation (HSCT) is a curative option for many children with cancer and certain genetic disorders. However, recipients of stem cell transplant must deal with years of disfigurement and symptoms arising from an undesirable side effect of transplant, specifically chronic graft-versus-host-disease (cGVHD).
* Children living with cGVHD often face many years of a disabling and painful chronic illness compounded by the side effects of prolonged immunosuppression, particularly long-term steroid use.
* Chronic GVHD can involve almost every organ although it most commonly affects the skin, eyes, mouth, liver, intestines, lung and the musculoskeletal system.
* There has been a large effort through the NIH cGVHD Consensus Consortium to standardize definitions, grading and response criteria for patients with cGVHD on clinical trials. Because of the absence of evidence suggesting which response criteria truly correlates with improvement, the NIH Consensus Panel has recommended following not only physical signs of chronic GVHD, but also symptoms of GVHD.
* The Lee cGVHD Symptom Score has been recognized as a core cGVHD outcome measure in the adult population, however, the instrument has not been validated for use in children/adolescents younger than 18, and many of the symptom terms used in the Lee cGVHD Symptom Scale may not be well understood by younger children.
* There is currently no available pediatric patient-reported outcome (PRO) measure of cGVHD symptom bother.

Primary Objective:

-To develop a psychometrically valid Pediatric cGVHD Symptom Scale (PCSS) and a companion caregiver-proxy measure as counterparts to the Lee cGVHD Symptom Scale.

Eligibility:

* Children 5 to 17 years of age for Project 1 or 8-17 years of age for Project 2, who have undergone prior allogeneic stem cell transplant
* Clinical diagnosis of cGVHD
* Currently receiving systemic treatment for cGVHD (including phototherapies), or has tapered systemic therapy for cGVHD to discontinuation within the past 12 months
* No evidence of malignant disease relapse including molecular relapse and minimal residual disease. Patients with mixed chimerism are eligible to participate
* Comprehend and speak English
* Caregivers of children 5-17 years of age with cGVHD enrolled as a proxies

Design:

* This multicenter non-interventional psychosocial trial will address the study aims in two projects: 1) a qualitative project using cognitive interviewing to confirm the comprehension and ease of response to the PCSS, and 2) a quantitative project to evaluate test-retest reliability, construct validity and responsiveness of the PCSS, as well as to explore concordance of symptom ratings by patients and caregiver proxies.
* In Project 1 (COMPLETE), we will conduct at least 20 cognitive interviews of patient and proxy dyads (caregiver) within each age group (5-7; 8-12; 13-17) for a sample of up to 90 pediatric transplant survivors with cGVHD to refine the symptom items and response choices to ensure that they resonate across the developmental spectrum. Cognitive interviews will evaluate the clarity and comprehension of the PCSS items, the ease and accuracy of judgement of the response choices, and any errors in understanding the response choices, and will refine the PCSS in accordance with study data, before proceeding to Project 2.
* In Project 2, we will evaluate test-retest reliability, construct validity, and responsiveness of the PCSS, in association with the NIH Global cGVHD Symptom Severity Score, the Peds QL, clinician ratings of organ specific cGVHD severity scores and cGVHD severity using the NIH criteria, in a sample of 100 pediatric transplant survivors with cGVHD reflecting two age groups (8-12 years; 13-17 years) of equal numbers and 20 caregivers of children age 5-7 who will serve as proxies. In participants ages 13-17, we will also compare responses on the PCSS with those from the Lee Scale, to determine the youngest age at which adolescent respondents can comprehend the Lee Scale.
* The overall accrual ceiling is 420, which includes pediatric and caregiver participants and accounts for inevaluable participants
* This study will include CCR investigators as well as extramural investigators at national and international study sites.

ELIGIBILITY:
* INCLUSION CRITERIA:

Pediatric Participant Inclusion Criteria:

* Children aged 5 to 17 years old (Project 1) or children aged 8 to 17 years old (Project 2)
* Clinical diagnosis of cGVHD following allogeneic stem cell transplant
* Currently receiving systemic treatment for GVHD (including phototherapies), or has had systemic therapy for GVHD tapered to discontinuation within the past 12 months
* No evidence of malignant disease relapse including molecular relapse and minimal residual disease. Patients with mixed chimerism are eligible to participate
* Must have an eligible caregiver proxy who is willing to participate in the study.
* Parent or guardian ability and willingness to sign a written informed consent document
* Must be able to comprehend and speak the English language
* Participants may enroll in both Project 1 and Project 2 of the study. Participation in Project 1 is not required in order to be eligible to participate in Project 2.

Caregiver Proxy Inclusion Criteria

* Adult (>=18 years old) caregiver of a child participating in Project 1 or Project 2; OR Adult (>=18 years old) caregiver of a child aged 5 to 7 years old who meets all Pediatric Participant Inclusion Criteria except Project 2 criteria noted above in the section Pediatric Participant Inclusion Criteria
* Must be willing and able to provide informed consent
* Must be able to comprehend and speak the English language

EXCLUSOIN CRITERIA:

Children may be excluded from this study if in the judgment of the Principal or Associate Investigator, the child is too ill, or the child s cognitive ability would compromise their ability to participate in study related procedures.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children of 5 to 17 years of age and their caregiver, who have undergone prior allogeneic stem cell transplant
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasability | 3 years
  To develop a psychometrically valid Pediatric cGVHD Symptom Scale (PCSS) and a companion parent-proxy measure as counterparts to the Lee cGVHD Symptom Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lori S Wiener, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (13):
- United States (12):
  - Children's Hospital Colorado (CHCO), Aurora, Colorado
  - Children s National Medical Center (CNMC), Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston Hospital, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital (JHH), Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - University of Pittsburgh - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children s Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital (TCH)-Baylor, Houston, Texas
  - The University of Texas MD Anderson Cancer Institute, Houston, Texas
  - Fred Hutchinson Cancer Center (FHCC), Seattle, Washington
- Children's & Women's Health Centre of British Columbia (CWHC of BC), Vancouver BC, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Derived] Mitchell SA, Hunter R, Fry A, Pavletic SZ, Widemann BC, Wiener L. Development and psychometric testing of a pediatric chronic graft-versus-host disease symptom scale: protocol for a two-phase, mixed methods study. Front Psychol. 2024 Jan 8;14:1243005. doi: 10.3389/fpsyg.2023.1243005. eCollection 2023. PMID 38259542
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0131.html